CLINICAL TRIAL: NCT03213028
Title: Family Planning Service Delivery Integration For HIV Positive And At-Risk Women In Botswana: A Hybrid Type 2 Clinical Intervention And Implementation Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of Botswana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 823794
Record Dates: First submitted 2017-05-03; First posted 2017-07-11 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Family Planning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Full group (Other): Our goal is to assess the feasibility and acceptability of incorporating family planning (FP) service delivery, using a program validated by the World Health Organization (WHO), into the established Cervical Cancer Prevention (CCP) programs of Botswana.
  Interventions: Other: WHO Decision-Making Tool for Family Planning Clients and Providers

INTERVENTIONS:
Other: WHO Decision-Making Tool for Family Planning Clients and Providers — Contraception decision-making tool

SUMMARY:
The goal of this pilot study is to assess both implementation outcomes (acceptability, feasibility and adoption) and clinical efficacy (contraceptive method uptake by women wishing to avoid pregnancy) using a Hybrid Type 2 study design of a family planning program being piloted by the Cervical Cancer Prevention Program in Gabarone, Botswana.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. English or Setswana speaking
3. Receiving CCP services at the clinic
4. 18-45 years of age
5. Able to give informed consent to study procedures, as determined by research/clinic staff

Exclusion Criteria:

1. Pregnant

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 248 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Provider acceptability rating | 6 months
  Likert scale 1-5, rating acceptability of offering family planning in this clinical setting.
Provider rating of feasibility | 6 months
  Likert scale 1-5, rating feasibility of offering family planning in this clinical setting
Provider report of adoption of the intervention | 6 months
  Comparing number of family planning methods offered by a provider pre- and post-intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Marina Hospital, Gabarone, Botswana

IPD SHARING:
Plan to Share IPD: No